CLINICAL TRIAL: NCT03094845
Title: Assessment of Safety and Clinical Tolerability of hdmASIT+TM Administered Subcutaneously in House Dust Mite-induced Allergic Rhinoconjunctivitis Patients
Brief Title: Safety and Clinical Tolerability of hdmASIT+TM Peptides Administered in HDM-induced Allergic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ASIT Biotech S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABT-hdmASIT001; 2016-000557-13 (EudraCT Number)
Record Dates: First submitted 2017-03-17; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: House Dust Mite Allergy
MeSH Terms: conditions — Dust Mite Allergy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo solution
- hdmASIT+TM (Experimental)
  Interventions: Biological: hdmASIT+TM

INTERVENTIONS:
Biological: Placebo solution — 15 injections over 7 weeks
  Arms: Placebo
Biological: hdmASIT+TM — 15 injections over 7 weeks
  Arms: hdmASIT+TM

SUMMARY:
hdmASIT+TM product is based on highly purified allergen fragments from house dust mites. The purpose of this study is to assess the safety and clinical tolerability of subcutaneous immunotherapy with hdmASIT+TM in patients with house dust mite-induced allergic rhinoconjunctivitis compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* A medical history of moderate to severe allergic rhinoconjunctivitis for house dust mite for at least 12 months (definition of allergy severity according to ARIA (Bousquet et al., 2001))
* A positive skin prick test to house dust mite Dermatophagoides pteronyssinus
* Specific IgE against house dust mite Dermatophagoides pteronyssinus ≥ 0.7 kU/L
* Positive response to Conjunctival Provocation Test (CPT)
* Being treated with anti-allergic medication for at least 12 months prior to enrollment
* For asthmatic patients: confirmed diagnosis of controlled asthma according to Global Initiative for Asthma (GINA) guidelines (steps 1-3, GINA 2014), FEV1 ≥ 80% of the patient's reference value

Exclusion Criteria:

* Previous immunotherapy with house dust mite allergens within the last 5 years
* Ongoing immunotherapy with house dust mite allergens or any other allergens
* History of severe systemic reactions and/or anaphylaxis, including to food (e.g. peanut, marine animals) or to Hymenoptera venom (e.g. bee, wasp stings) or to medication (e.g. penicillin), etc.
* Partly controlled or uncontrolled asthma according to GINA guidelines (GINA 2014)
* Chronic asthma or emphysema, particularly with a forced expiratory volume in 1 second (FEV1) < 80% of the patient's reference value (ECSC)
* History of a respiratory tract infection and/or exacerbation of asthma within 4 weeks before the screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-23 (Actual)

PRIMARY OUTCOMES:
Solicited adverse events | up to 7 weeks
  * Local reactions at the injection site
  * Allergic systemic reactions

SECONDARY OUTCOMES:
Unsolicited adverse events and serious adverse events (SAEs) | up to 12 weeks
Physical examinations (body systems) and vital signs (heart rate, systolic and diastolic blood pressure) | up to 12 weeks
Laboratory investigations (haematology, clinical biochemistry, immunological parameters) | up to 12 weeks
Pulmonary functions (FEV1) for asthmatic patients | up to 7 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Carl Gustav Carus, Dresden, Germany